CLINICAL TRIAL: NCT02195674
Title: Exploring Massage Benefits for Arthritis of the Knee (EMBARK): Post-study Massage Questionnaire
Brief Title: EMBARK Follow-up Project
Acronym: EFP
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00054004; 3R01AT004623-06S2 (NIH)
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the EMBARK Follow-up Project (EFP) is to determine if there is a significant correlation between post-study massage-seeking and changes in pain reported by participants during the Exploring Massage Benefits for Osteoarthritis of the Knee (EMBARK) parent study (NCT00970008). The EFP hypothesizes that a positive correlation exists between pain relief during the parent study and post-study massage-seeking behavior.

ELIGIBILITY:
Inclusion Criteria:

* Completed in the EMBARK parent study.

Exclusion Criteria:

* Did not complete the EMBARK parent study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the EMBARK parent study.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
EMBARK Follow-up Project Questionnaire (EFPQ) | Eight weeks
  The EFPQ is an original set of questions, designed and validated by Dr. Jerger under the supervision of NCCAM and Dr. Ruth Wolever to be administered by email or phone to address the specific aims of this project.

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Perlman, MD, MPH, Principal Investigator — Duke University